CLINICAL TRIAL: NCT05974202
Title: Augmenting Cognitive-behavioral Therapy With rTMS of the Medial Prefrontal and Anterior Cingulate Cortices for the Treatment of Cocaine Use Disorder
Brief Title: rTMS and Cognitive-behavioral Therapy for Cocaine Use Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Columbia University (Other)
Responsible Party: Principal Investigator, John Mariani MD, Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UG3DA056138 (NIH)
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Cocaine Use; Cocaine Dependence; Cocaine Use Disorder; Cocaine Use Disorder, Moderate; Cocaine Use Disorder, Severe
Keywords: Repetitive transcranial magnetic stimulation; rTMS; TMS; Cognitive behavioral therapy; CBT; Functional magnetic resonance imaging; fMRI
MeSH Terms: conditions — Cocaine-Related Disorders; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Active high-frequency stimulation vs. sham (placebo) stimulation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active (high-frequency) rTMS (Active Comparator): Daily high-frequency (10 Hz) repetitive transcranial magnetic brain stimulation for 3 weeks (15 sessions).
  Interventions: Device: Active H7-coil repetitive transcranial magnetic stimulation (rTMS)
- Sham (placebo) rTMS (Placebo Comparator): Sham rTMS uses the same device and mimics the auditory and scalp sensations without stimulating the brain.
  Interventions: Device: Sham H7-coil repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: Active H7-coil repetitive transcranial magnetic stimulation (rTMS) — A magnetic current created by the device creates an electrical current in the brain to stimulate the medial prefrontal cortex and dorsal anterior cingulate cortex.
  Arms: Active (high-frequency) rTMS
Device: Sham H7-coil repetitive transcranial magnetic stimulation (rTMS) — A sham coil is in the same helmet as the active coil. The sham coil mimics the sound, scalp sensations, and facial muscle activation caused by the active coil, but does not create an electrical current in the brain.
  Arms: Sham (placebo) rTMS

SUMMARY:
The goal of this clinical trial is to compare the effects of active repetitive transcranial magnetic stimulation (rTMS) to sham (placebo) rTMS prior to cognitive-behavioral therapy (CBT) as a treatment for adults with cocaine use disorder. The main questions it aims to answer are:

* Is rTMS safe and feasible as an augmentation for CBT for the treatment of cocaine use disorder?
* What is the brain mechanism of rTMS?
* Will active rTMS (compared to sham rTMS) followed by CBT help adults with cocaine use disorder achieve abstinence from cocaine?

Participants will:

* Have two brain MRI scans;
* Undergo 3 weeks of daily rTMS (or sham) treatments (15 sessions), and;
* Have 12 weeks of once-weekly cognitive-behavioral therapy for the treatment of cocaine use disorder.

Researchers will compare active (real) rTMS to sham (placebo) rTMS. All participants will receive cognitive-behavioral therapy.

The former principle investigator, Dr. Derek Blevins, has vacated his position (February 2025), and has transferred the principle investigator role to Dr. John Mariani, the STARS Clinic Director.

DETAILED DESCRIPTION:
Cocaine use disorder (CUD) remains a significant public health problem given that many patients fail to respond to existing therapies (Dutra et al., 2008). Treatment refractory CUD may be explained, in part, by abnormal neurocircuitry. The medial prefrontal cortex (mPFC) and dorsal anterior cingulate cortex (dACC) have demonstrated altered functioning in CUD (Hanlon et al., 2016). Compared to controls, participants with CUD show consistent changes to the mPFC/dACC, including hypoactivation during cognitive and attentional tasks (Bolla et al., 2003; Kaufman et al., 2003; Kubler et al., 2005), hyperactivation during drug cue exposure (Garavan et al., 2000; Grant et al., 1996), and lower grey matter volumes (Ersche et al., 2011; Matochik et al., 2003).

Imaging studies also show that these alterations in the mPFC/dACC are associated with an impaired response to treatment. Hypoactivation of the mPFC/dACC region of the fronto-cingular network during the Color-Word Stroop task, a measure of cognitive interference and response inhibition, is associated with faster relapse rates (Brewer et al., 2008). Greater activation of the fronto-cingular network during incongruent stimuli on the Stroop task is also associated with poorer outcomes in CUD participants receiving cognitive behavioral therapy (CBT) (Worhunsky et al., 2013). When using the Drug Stroop task, better performance was associated with a longer duration of cocaine abstinence during CBT (DeVito et al., 2018). Thus, processing deficits across these brain regions likely contribute to the limited success of behavioral interventions for CUD, resulting in high dropout rates and a lack of treatment response.

Our goal is to target the mPFC/dACC with repetitive transcranial magnetic stimulation (rTMS) to investigate its impact on neurocognitive function and response to treatment in CUD. We will use the H7-coil, which targets the mPFC/dACC and has been FDA-cleared as a treatment for obsessive-compulsive disorder (Carmi et al., 2019). Previous work by our group showed that high-frequency (10 Hz) rTMS with the H7-coil led to a significant reduction in choices for cocaine in the human laboratory setting (Martinez et al., 2018). Additional studies using rTMS for CUD have targeted the dorsolateral or ventromedial PFC and demonstrated reduction in craving and drug cue reactivity (Ekhtiari et al., 2019; Antonelli et al., 2021; Kearney-Ramos et al., 2018; Kearney-Ramos et al., 2019).

Despite these promising findings, sham-controlled clinical trials investigating the effect of rTMS on abstinence and cocaine consumption are lacking. In this trial, our goal is to investigate rTMS as a potential treatment for CUD. Treatment-seeking volunteers with moderate/severe CUD will undergo three weeks (15 daily sessions) of outpatient, randomized, double-blinded, sham-controlled, high-frequency (10 Hz) rTMS to the mPFC/dACC with the H7-coil followed by standardized CBT. We will evaluate feasibility, safety, and the effect of rTMS on the mPFC/dACC using functional magnetic resonance imaging (fMRI) and clinical outcome measures (cocaine use). This outcome data will inform a larger clinical trial to evaluate rTMS as an augmentation for CBT outcomes in moderate/severe CUD and further explore the associated neural mechanisms of rTMS in this clinical population.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22-65;
2. Able to give informed consent and comply with study procedures;
3. Meets DSM-5 criteria for current moderate/severe CUD and are treatment-seeking;
4. Used cocaine at least 9 days in the past 28 days, with at least weekly cocaine use;
5. Agree to no more than moderate alcohol consumption (<15 drinks/week for men and <8 drinks/week for women) and to avoid using amphetamine/methamphetamine and non-prescribed benzodiazepines or barbiturates; and
6. Women of childbearing potential must agree to use a method of contraception with proven efficacy and agree to not become pregnant during the study.

Exclusion Criteria:

1. Meets DSM-5 criteria for current moderate/severe major depressive episode, OCD, bipolar disorder, schizophrenia or any psychotic disorder other than transient psychosis due to substance use;
2. Hamilton Depression Rating Scale score > 17;
3. Young Mania Rating Scale score >10;
4. Meets DSM-5 criteria for current moderate/severe other substance use disorder (aside from tobacco use disorder; physiologic dependence on any other substance other than nicotine, including alcohol, is exclusionary);
5. Heavy weekly alcohol drinking as defined by an average of >14 drinks/week for men or >7 drinks/week for women on average during the past 28 days;
6. Prior alcohol, benzodiazepine, or barbiturate withdrawal that resulted in hospitalization, medical detoxification, or resulted in seizures or delirium tremens;
7. More than twice weekly use of non-prescribed medications/drugs that may change the seizure threshold, including benzodiazepines, barbiturates, GHB/GBL, amphetamines/methamphetamine;
8. Any other current DSM-5 psychiatric disorder(s) that in the investigator's judgment are unstable, would be disrupted by study procedures, or are likely to require pharmacotherapy or psychotherapy during the study period;
9. Significant current suicide risk, indicated by either: (1) "yes" response on #3, 4, or #5 on the C-SSRS and a psychiatric risk assessment indicating a moderate or high risk of suicide or (2) suicidal behavior in the past 3 months (note: non-suicidal self-injurious behavior is not exclusionary);
10. Females with a positive urine pregnancy test;
11. Clinically significant abnormal cardiac functioning per electrocardiogram (ECG) (required for any participant age 60 years and older);
12. Seizure history including: seizure disorder/epilepsy, alcohol/drug withdrawal seizure, or seizure deemed by the study physician to be related to cocaine intoxication/withdrawal (note: febrile seizures are not exclusionary)
13. Other medical conditions that are relatively contraindicated with TMS (seizure disorders, glaucoma, increased intracranial pressure, severe migraines, stroke, brain lesions, pregnancy or breast-feeding, neurodegenerative disease, meningoencephalitis, intracerebral abscess, parenchymal or leptomeningeal cancers);
14. Medications that lower seizure threshold and in the opinion of the investigator impose significant seizure risk for the individual (including bupropion, antipsychotics, lithium, anticholinergics, and tricyclic antidepressants);
15. Cognitive disorder (MMSE <25);
16. Disqualifying response on the TMS Adult Safety Screen (TASS);
17. Implanted devices or stimulators (cardiac pacemakers, vagus nerve stimulators, spinal cord stimulators, cochlear implant);
18. Currently taking ototoxic medications (aminoglycosides, cisplatin);
19. Metal implants or paramagnetic objects in the body that prohibits MR scanning;
20. Claustrophobia that prohibits MR scanning; or
21. Legally mandated (e.g., to avoid incarceration or other penalties) to participate in SUD treatment program.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants receiving at least 10 out of 15 rTMS sessions | 3 weeks
  Feasibility will be measured as the total percentage of participants who receive the defined number of rTMS sessions
Number of participants in the active rTMS arm experiencing an rTMS-emergent adverse event | 3 weeks
  Safety of rTMS will be measured by the absolute number of serious adverse events that occur in the active rTMS arm
Percent change of medial prefrontal cortex and dorsal anterior cingulate cortex activity on fMRI during the Drug Stroop Task | 3 weeks
  Neural mechanism will be evaluated by comparing the active and sham rTMS groups during the fMRI task by comparing baseline fMRI and post-rTMS fMRI measures
Percentage of participants who achieve 3 weeks of abstinence during the final 12 weeks of the trial | 12 weeks
  Efficacy regarding cocaine use outcomes will be evaluated by comparing the active and sham rTMS groups during the final 12 weeks of the trial while the participants are receiving cognitive behavioral therapy. 3 weeks of consecutive abstinence is defined as: 1. No cocaine use is self-reported per timeline followback; 2. At least 6 urine drug screens are completed during the 3 weeks of continuous abstinence, and all are negative (with the exception of any positive urine in the first 4 days of the first week of the three weeks of self-reported abstinence, as urine may remain positive for up to 4 days after an episode of use), and; 3. At least 1 urine drug screen is completed each week during the 3 weeks of self-reported continuous abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: John Mariani, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute (NYSPI) / Substance Treatment and Research Service (STARS), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results published in this report (after de-identification) (text, tables, figures).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning twelve months and ending 5 years after article publication.
Access Criteria: To researcher who provides a methodologically sound proposal to achieve aims in approved proposal.